CLINICAL TRIAL: NCT02690688
Title: The Influence of Pneumoperitoneum and Open Abdominal Surgery on Dynamic Preload Variables
Brief Title: Intra-abdominal Pressure and Dynamic Preload Variables
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Luebeck (Other)
Responsible Party: Principal Investigator, Matthias Heringlake, Professor of Anesthesiology, Deputy Director Cardiac Anesthesia, Dept. of Anesthesiology and Intensive Care Medicine, University of Luebeck
Other Study IDs: HL-2016-Monitoring
Record Dates: First submitted 2016-02-18; First posted 2016-02-24 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-02

CONDITIONS: Pneumoperitoneum
Keywords: Pulse Pressure Variation; NIRS; Pneumoperitoneum; Abdominal surgery
MeSH Terms: conditions — Pneumoperitoneum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Pneumoperitoneum: Patients scheduled for laparoscopic (minimal invasive) abdominal surgery supported by pneumoperitoneum. Hemodynamic monitoring will be performed using Vigileo® monitor, Edwards Lifescience
  Interventions: Device: determination of dynamic preload variables
- Open Surgery: Patients scheduled for conventional (open) abdominal surgery. Hemodynamic monitoring will be performed using Vigileo® monitor, Edwards Lifescience
  Interventions: Device: determination of dynamic preload variables

INTERVENTIONS:
Device: determination of dynamic preload variables

SUMMARY:
Dynamic preload variables like pulse-pressure and stroke volume variation may be used to predict fluid responsiveness in patients during controlled ventilation. Previous work has shown that a rapid decrease in intra-abdominal pressure may lead to an increase in dynamic preload parameters, suggestive of a fluid deficit - despite fluid status had not changed [van Lavieren M 2014].

The results of this study are limited by the fact that a non-invasive and uncalibrated hemodynamic monitoring system (Nexfin™) was used.

The present study thus aims to evaluate the effects of abdominal pressure changes on dynamic preload parameters (PPV and SVV) employing conventional, invasive hemodynamic monitoring (Vigileo®, Edwards Lifescience) in open abdominal surgery as well as in minimal invasive surgical procedures with pneumoperitoneum.

DETAILED DESCRIPTION:
Hemodynamic monitoring is an essential part of modern anesthesia. Establishing and maintaining normovolemia during surgery is of high clinical relevance. Various studies suggest that dynamic preload parameters like stroke volume variation (SVV) and pulse pressure variation (PVV) are superior for interpretation and management of fluid status than static parameters like central venous pressure (CVP). Consequently, dynamic preload parameters have been integrated in recent guidelines for hemodynamic and fluid management.

Animal studies have shown reliable results for SVV and PVV to discriminate fluid-responder from non-responders if intraabdominal pressure is increased [Jacques D 2011]. In contrast to these findings, van Lavieren and colleagues have shown an inappropriate increase in measured dynamic preload parameters upon opening the abdomen using a non-invasive and uncalibrated system (Nexfin™). The present study thus aims to determine the effects of changes in abdominal pressure on dynamic preload parameters (PPV and SVV) (primary objective) employing an established invasive hemodynamic monitoring tool (Vigileo®, Edwards Lifescience) during open abdominal surgery as well as in minimal invasive surgical procedures using pneumoperitoneum.

Secondary objective is the effect of changes of cerebral oximetry readings during open and laparoscopic procedures and their relation to changes in cardiac index.

Elective ASA I-III patients scheduled for open and laparoscopic abdominal surgery will be enrolled according the planned operative procedure (open abdominal surgery or minimal invasive surgical procedures using pneumoperitoneum) and assignment. 60 patients (30/group) will be included according to a sample size calculation based on the data by van Lavieren.

Prior to induction of anesthesia an invasive blood pressure monitoring (radial artery) will be established and connected to a Vigileo® monitor (Edwards Lifescience). Additionally, bilateral optodes for the monitoring of cerebral oxygenation will be applied (INVOS, Somanetics). Ventilation, anesthesia and fluid management will be standardized.

Hemodynamic variables will be recorded prior to induction of anesthesia, after anesthesia was induced, and at the initial time point of pneumoperitoneum/open abdomen.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III patient
* Signed agreement
* Surgical procedure with open abdomen surgery or pneumperitoneum
* Age > 18 Years
* Intubation

Exclusion Criteria:

* BMI ≥ 35 kg/m2
* Need for catecholamines
* Cardiac arrhythmia
* Fluid resuscitation during measurements
* Ongoing periduralcatheter-therapy
* Missing agreement
* Disposition for MH
* Inclusion in other investigations < 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with the need of an abdominal operation. According operation technique patients gets assigned to one of the groups.
  In- and exculsion criteria are given below.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2016-03; Primary Completion 2017-03 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Influence of pneumoperitoneum or open abdominal surgery on dynamic preload parameters | Mesurements during one minute after induction of pneumoperitoneum or open abdominal surgery

SECONDARY OUTCOMES:
Influence of pneumoperitoneum or open abdominal surgery on cerebral oxymetry | Mesurements during one minute after induction of pneumoperitoneum or open abdominal surgery
Correlation of cerebral oxymetry and cadiac index in pneumoperitoneum or open abdominal surgery | Mesurements during one minute after induction of pneumoperitoneum or open abdominal surgery

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Heringlake, MD, Principal Investigator — Professor of Anesthesiology, Deputy Director Cardiac Anesthesia, Dept. of Anesthesiology University of Lübeck, Ratzeburger Allee 160, 23538 Lübeck
Locations (1):
- Department of Anesthesiology, University of Luebeck, Lübeck, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] van Lavieren M, Veelenturf J, Hofhuizen C, van der Kolk M, van der Hoeven J, Pickkers P, Lemson J, Lansdorp B. Dynamic preload indicators decrease when the abdomen is opened. BMC Anesthesiol. 2014 Oct 14;14:90. doi: 10.1186/1471-2253-14-90. eCollection 2014. PMID 25337036
- [Background] Jacques D, Bendjelid K, Duperret S, Colling J, Piriou V, Viale JP. Pulse pressure variation and stroke volume variation during increased intra-abdominal pressure: an experimental study. Crit Care. 2011;15(1):R33. doi: 10.1186/cc9980. Epub 2011 Jan 19. PMID 21247472